CLINICAL TRIAL: NCT05465447
Title: The Long-term Outcome After Cataract Surgery With Toric Intraocular Lens Implantation
Brief Title: The Long-term Outcome After Toric Intraocular Lens Implantation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Other Study IDs: TORIC-long term
Record Dates: First submitted 2022-06-20; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Corneal Astigmatism; Cataract
MeSH Terms: conditions — Astigmatism; Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Toric IOL: This study included the patients who underwent cataract surgery with the toric IOL(SN6ATX) implantation. Preoperative and postoperative corneal astigmatism, short-term and long-term postoperative total astigmatism were the main outcome indicators. Preoperative corneal astigmatism (Pentacam and IOLMaster) would be obtained from outpatient and inpatient medical records, and the IOL axis should be calculated before surgery. Short-term postoperative (1-3 months) subjective optometry results; Long-term postoperative (3-5 years) corneal astigmatism (Pentacam and IOLMaster), subjective optometry results, and axial lens would be observed using SSOCT after pupil dilation.
  Interventions: Device: subjective refraction

INTERVENTIONS:
Device: subjective refraction — Short-term postoperative (1-3 months) and long-term postoperative (3-5 years) subjective optometry results were measured by subjective refraction.

SUMMARY:
Corneal astigmatism is refractive error that impairs uncorrected visual acuity. When patients undergo cataract surgery, implantation of toric IOL is deemed the most effective choice for correcting corneal astigmatism and reducing postoperative spectacle dependence. Previous studies report that the visual effects and rotational stability of toric IOLs are well maintained over 1- or 2-year follow-up periods. However, the long-term changes in the effects of toric IOLs remain unclear.

DETAILED DESCRIPTION:
Corneal astigmatism is refractive error that impairs uncorrected visual acuity. When patients undergo cataract surgery, implantation of toric IOL is deemed the most effective choice for correcting corneal astigmatism and reducing postoperative spectacle dependence. Previous studies report that the visual effects and rotational stability of toric IOLs are well maintained over 1- or 2-year follow-up periods. However, there is a long-term against-the-rule (ATR) change of corneal astigmatism with aging，which influences the long-term outcomes of refractive surgery. The long-term changes in the effects of toric IOLs remain unclear. This study aim to observe the clinical effect of Toric IOL implantation in the correction of corneal astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* ≥18years old
* Regular astigmatism
* Corneal astigmatism ≥ 0.75D

Exclusion Criteria:

* Macular degeneration and retinal disease, history of glaucoma, corneal disease
* Previous corneal or intraocular surgery, and history of ocular inflammation.
* Pupils can not be dilated (< 7mm)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From December 2012 to present, cataract patients underwent phacoemulsification combined with Toric IOL(SN6ATX) implantation by an experienced ophthalmologist (Dr. Zhao Yune) in Wenzhou Medical University Affiliated Eye Hospital(hangzhou branch).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
changes of magnitude of corneal astigmatism from pre-surgery to 3-5 years after surgery | before surgery and 3-5 years after surgery
  using Pentacam measure cornea astigmatism of the subjects
changes of axis of corneal astigmatism from pre-surgery to 3-5 years after surgery | before surgery and 3-5 years after surgery
  using Pentacam measure cornea astigmatism of the subjects
changes of manifest refractive astigmatism from1 -3 months after surgery to 3-5 years after surgery | 1-3 months after surgery and 3-5 years after surgery
  measured using subjective refraction by Professional optometrists